CLINICAL TRIAL: NCT03995498
Title: Individualized Carbohydrate Intake Strategy to Improve Blood Glucose Control During Team Sports in Children and Adolescents With Type 1 Diabetes: A Carowanis Camp Study
Brief Title: Individualized Carbohydrate Intake Strategy to Improve Blood Glucose Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Full professor, Institut de Recherches Cliniques de Montreal
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SNACK-camp
Record Dates: First submitted 2019-06-20; First posted 2019-06-24 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Type 1 Diabetes
Keywords: Exercise; Physical activity; Carbohydrates; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity; Hypoglycemia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized carbohydrate intake (Active Comparator): Based on glucose sensor level, carbohydrate (orange juice, Oasis classic) will then be given as follow:
  If sensor glucose level is under < 4.5 mmol/L, the camp staff will treat hypoglycemia according to the camp procedure, If sensor glucose level is between 4.5 and 7.0 mol/L, 0.5g of CHO/kg body weight will be given, If sensor glucose level is between 7.1 and 10.0 mmol/L, 0.25g of CHO/kg body weight will be given, If sensor glucose level is between 10.1 and 15.0 mmol/L, no CHO will be given, If sensor glucose level is > 15.1 mmol/L, the camp staff will treat hyperglycemia according to the camp procedure.
  Interventions: Other: Physical activity; Other: FreeStyle Libre; Other: SenseWear Armband
- Usual camp protocol (Active Comparator): As per camp routine care, there will be no mandatory glucose level measurement before the start of physical activity if no symptoms of hypoglycemia or hyperglycemia appear.
  Interventions: Other: Physical activity; Other: FreeStyle Libre; Other: SenseWear Armband

INTERVENTIONS:
Other: Physical activity — Participants will engage in team sports exercise twice a day: from 9h:30 to 10h:30 and from 11h:00 to 12h:00.
Other: FreeStyle Libre — Glucose levels will be measured by the FreeStyle Libre
Other: SenseWear Armband — Energy expenditure during physical activity sessions will be measured with the SenseWear Armband.

SUMMARY:
The objective of this study is to test whether an individualized carbohydrate intake based on weight and pre physical activity glucose level is more effective than usual camp care to improve glucose control in children and adolescents engaging in team sports (basketball, soccer, hockey) during a summer camp.

At the enrollment interview, in addition to collecting patient's information (age, sex, diabetes duration, recent A1c, type of treatment, insulin doses body weight, concomitant diseases, diabetes complications and history of severe hypoglycemia), a continuous glucose monitoring system (FreeStyle Libre) will be installed by a nurse. At least, eight sports sessions per participant are planned for this study. In a randomized order, the individualized carbohydrate intake will be applied during at least 4 interventions sport sessions while at least 4 with matching types of sports will be used as control sessions. Two sport sessions are routinely scheduled at the camp each day; from 9h:30 to 10h:30 and from 11h:00 to 12h:00. For intervention sessions that involve individualized carbohydrate intake, the FreeStyle Libre will be scanned 0-10 minutes before the start of the team sport. Carbohydrates will then be given in the amount of 0.5g/kg for glucose levels between 4.5 to 7.0 mmol/L and 0.25g/kg for glucose levels between 7.1 to 10.0 mmol/L and none will be given if glucose levels are between 10.1 and 15.0 mmol/L. When glucose levels are below 4.5 mmol/L or above 15.0 mmol/L, the camp staff will take care of hypoglycemia/hyperglycemia treatment. During control sessions, as per camp routine care, there will be no measurement of glucose levels before the start of physical activity.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the 7 and 16 years of old.
2. Clinical diagnosis of type 1 diabetes for at least 6 months.
3. Using continuous subcutaneous insulin infusion therapy or multiple daily injections.
4. HbA1c ≤ 12.0%.
5. Practicing team sports (soccer, basketball, hockey, tennis) at the summer camp.

Exclusion Criteria:

1. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
2. Severe hypoglycemic episode within two weeks of inclusion in the study.
3. Using the Medtronic 670G Insulin Pump as a treatment Mode
4. Current use of oral glucocorticoid medication (except low stable dose according to investigator judgement). Stable doses of inhaled steroids are acceptable.
5. Acute disease in the last 3 months that would affect ability to do physical activity.
6. Other serious medical illness likely to interfere with study participation or with the ability to complete the exercise periods by the judgment of the investigator (e.g. orthopedic limitation).

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Percentage of time of interstitial glucose concentrations spent between 4.0-10.0 mmol/L | 60 minutes

SECONDARY OUTCOMES:
Change in glucose concentrations | 60 minutes
Mean time (minutes) to the first hypoglycemic event | 60 minutes
Mean interstitial glucose concentration | 60 minutes
Standard deviation of glucose concentration | 60 minutes
Percentage of time of interstitial glucose concentrations spent below 4.0 mmol/L | 120 minutes
Percentage of time of interstitial glucose concentrations spent above 10.0 mmol/L | 120 minutes
Number of participants with an exercise-induced hypoglycemia below 4.0 mmol/L | 120 minutes
Number of participants with an exercise-induced hypoglycemia below 3.5 mmol/L | 120 minutes
Total number of confirmed hypoglycemia episodes requiring treatment | 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Montreal Clinical Research Institute
Locations (1):
- Montreal Clinical Research Institute, Montreal, Quebec, Canada